CLINICAL TRIAL: NCT07083336
Title: Liver Fat as a Dietary Target of the Chinese Medical Nutrition Therapy (CMNT) Diet for Treating Type 2 Diabetes With Nonalcoholic Fatty Liver Disease
Brief Title: Liver Fat as a Dietary Target of the Chinese Medical Nutrition Therapy (CMNT) Diet for Treating Type 2 Diabetes With Nonalcoholic Fatty Liver Disease (Version 3.0)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State Key Laboratory of Subhealth Intervention Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 3.0
Record Dates: First submitted 2025-07-08; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus; Metabolic Dysfunction-associated Steatotic Liver Disease
Keywords: Comorbid MASLD and T2DM; Intermittent energy restriction
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: CMNT diet (Experimental): The CMNT group was instructed to consumed the provided CMNT diet consisting of 6 cycles of 5 consecutive days followed by 10 days of ad libitum food consumption. Participants received a 917 kcal/day preprepared human CMNT diet (44.75% carbohydrate, 9.1% protein and 46.15% fat) for 5 consecutive days per cycle
  Interventions: Other: CMNT diet
- Usual Care (No Intervention): Dietary recommendations based on the Guideline for the prevention and treatment of type 2 diabetes mellitus in China (2020 edition) as the control group

INTERVENTIONS:
Other: CMNT diet — Hypocaloric CMNT diet plan: A diet plan with intermittent use of enriched traditional-Chinese-medicinal-foods CMNT diet
  Arms: Experimental: CMNT diet

SUMMARY:
This study aims to explore the efficacy of CMNT, an intermittent energy restriction (iER) intervention, in managing Chinese adults with type 2 diabetes and non-alcoholic fatty liver disease. An interim analysis will be added to the planned 120-participant CMNT intervention program to compare intervention efficacy with the usual care control group and assess potential risks associated with dietary interventions.

DETAILED DESCRIPTION:
Study Protocol Amendments (v3.0) are as follows:

1. Addition of Interim Analysis. Rationale: The purpose of adding an interim analysis is to evaluate the effectiveness of the CMNT dietary intervention during this clinical trial, while also assessing participant compliance and the safety of the energy-restricted diet.
2. Expansion of BMI Inclusion Criteria. The BMI inclusion criterion was revised from "18-35" to " > 18" (removing the upper limit) to include patients with higher BMI values. Rationale: In clinical practice, some patients with a BMI over 35 have shown interest in participating in this study. After evaluation by physicians, these patients can be included.
3. Increase in the Number of Multicenter Sites. The number of centers increased from 3 to 6. Rationale: Expanding the number of multicenter sites accelerates participant recruitment. Given the study's focus on patients with T2D and NAFLD, the recruitment of patients with comorbidities is relatively challenging. Additionally, expanding the number of centers enhances the generalizability of the study's conclusions, making them applicable to patients in more regions.
4. Clarification and Revision of Secondary Objectives and Corresponding Evaluation Criteria. Addition of metabolomics content to identify key metabolites in CMNT intervention; Screening for key microbial taxa post - CMNT intervention based on gut microbiota results; Validation of the causal relationship between diet and gut microbiota using fecal transplantation; Rationale: Incorporating gut microbiota and metabolomics indicators helps better explore the mechanism of CMNT dietary intervention in this population.
5. The participant recruitment period has been extended to May 5, 2026. Rationale: Due to the severe COVID-19 pandemic during 2022-2023, coupled with the fact that this study focuses on comorbidities, the number of eligible participants has been significantly lower compared to studies involving general T2D patients. Furthermore, as most individuals currently do not prioritize fatty liver screening, participant recruitment has progressed more slowly than anticipated. Therefore, an extension of the recruitment period is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes and NAFLD.
* Age between 18 and 75 years.
* Body mass index (BMI) > 18.0 kg/m2
* Weight stable for at least 3 months prior to the study (gain or loss <4kg).
* Stable treatment for at least 3 months with 1-3 oral
* antidiabetic medications (with or without insulin therapy), or not yet receiving antidiabetic medication prior to the beginning of the study.
* Able to give written informed consent.

Exclusion Criteria:

* Participants meeting any of the following criteria will not be allowed to participate in the trial:
* Use of any of the following medications or treatments:
* Use of other medications that may affect glucose metabolism within the past 2 months, including systemic glucocorticoids (excluding inhaled or topical use), growth hormones, etc.;
* Use of antihypertensive or lipid-lowering medications that have not reached a stable dosage before screening;
* Presence of any of the following medical histories or conditions:
* History or presence of any cardiac disease within the past 6 months;
* Decompensated heart failure (NYHA Class III or IV);
* Unstable angina, myocardial infarction, coronary artery bypass grafting, or coronary stenting;
* Uncontrolled or severe arrhythmias (e.g., long QT syndrome), as assessed by the investigator as unsuitable for trial participation;
* History of hemorrhagic or ischemic stroke within the past 6 months, as assessed by the investigator as unsuitable for trial participation;
* Medical history of cerebral thrombosis, cerebral vascular blockage, encephalic angioma, transient ischemic attack, cerebral hemorrhage, stroke, hydrocephalus, or malignant brain tumor;
* History of carotid artery stenting;
* Urinary system conditions such as nephrotic syndrome, uremia, polycystic kidney disease, kidney transplantation, unilateral nephrectomy/congenital solitary kidney, renal atrophy, renal tumor;
* Digestive system conditions such as ascites, liver cirrhosis, liver fluke infection, severe hepatitis, gastric varices;
* Nervous system conditions such as cerebellar atrophy, demyelinating diseases, cerebral palsy, Parkinson's disease, mania, schizophrenia;
* Respiratory system conditions such as pulmonary embolism, cor pulmonale;
* Musculoskeletal system conditions such as arterial rupture, myeloma;
* Immune system conditions such as Behçet's disease, lupus erythematosus;
* Conditions such as chondrosarcoma, liposarcoma, brucellosis, leukemia;
* History of malignant tumor within the past 5 years, or currently under evaluation for potential malignancy;
* History of unstable or treatment-requiring proliferative retinopathy or macular edema within the past 6 months;
* History of diabetic ketoacidosis or hyperosmolar nonketotic diabetic coma within the past 6 months;
* Currently suffering from lower extremity arteriosclerotic occlusive disease; History of severe infection or severe trauma within the past 1 month;
* History of ≥2 severe hypoglycemic episodes within the past year;
* Currently suffering from clinically significant urinary tract/genital infection, or a history of complicated urinary tract infections, or recurrent urinary tract infections within the past 6 months;
* Currently suffering from uncontrolled hypertension, defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg at screening/baseline, or systolic blood pressure ≤90 mmHg and/or diastolic blood pressure ≤60 mmHg;
* Currently suffering from uncontrolled thyroid dysfunction;
* History of other severe endocrine diseases, such as multiple endocrine neoplasia;
* History of severe hepatic or renal disease;
* Suspected or confirmed history of alcohol or drug abuse;
* Blood donation or blood loss ≥400 mL within the past 3 months;
* Presence of severe psychiatric disorders or language barriers, unwillingness or inability to fully understand and cooperate;
* Pregnant or breastfeeding women;
* Any other conditions deemed unsuitable for trial participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Controlled attenuation parameter (CAP) value by transient elastography | 3, 6, 12, 24 months
  The CAP score, which be measured by FibroScan, will be used to quantify and detect liver fat. CAP < 238 dB/m indicated no hepatic steatosis, 238 ≤ CAP ≤ 259 dB/m denoted mild steatosis, 260 ≤ CAP ≤291 dB/m indicated moderate steatosis, and CAP > 291 dB/m denoted severe steatosis.
HbA1C | 3, 6, 12, 24 months
  Blood test to measure glucose control

SECONDARY OUTCOMES:
γ-GGT | 3, 6, 12, 24 months
  γ-glutamyl transferase (γ-GGT) will be assessed for liver function tests
Body Mass Index (BMI) | 3, 6, 12, 24 months
  Body Mass Index (BMI) will be measured as an anthropometric parameter (kg/m²)
Fasting blood glucose | 3, 6, 12, 24 months
  Fasting blood glucose (mmol/L) will be assessed among Glycemic Homeostasis Parameters
Fasting insulin | 3, 6, 12, 24 months
  Fasting insulin (μIU/mL) will be assessed among Glycemic Homeostasis Parameters
Blood lipid | 3, 6, 12, 24 months
  triglyceride, total cholesterol, low-density lipoprotein cholesterol (LDL-C) and high-density lipoprotein-cholesterol (HDL-C)
Liver fibrosis markers | 3, 6, 12, 24 months
  Liver stiffness measurement (LSM) value by transient elastography DiabetesLiver score Fibrotic non-alcoholic steatohepatitis index (FNI) Fibrosis-4 index (FIB-4) NAFLD fibrosis score (NFS)
Hepatic steatosis Markers | 3, 6, 12, 24 months
  Fatty liver index (FLI) Hepatic steatosis index (HSI)
Food Frequency Questionnaire (FFQ) | 3, 6, 12, 24 months
  The Food Frequency Questionnaire (FFQ) typically estimates nutrient intake based on food consumption frequency, with a common range of 800-5000 kcal/day for adults.
Metabolomics | 3, 6, 12, 24 months
  Concentration of Key Serum Metabolites Identified by Metabolomics Before and After CMNT Intervention in All Participants
Gut microbiota | 3, 6, 12, 24 months
  Change in Gut Microbiota Composition (Relative Abundance at species Level) Before and After CMNT Intervention in All Participants

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Physical Examination Center of Gezhouba central hospital of Sinopharm, Yichang, Hubei
  - Hunan Shanshui physical examination center, Changsha, Hunan
  - Jinheyuan Outpatient Department, National Sub-health Intervention Technology Achievement Application Center, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No